CLINICAL TRIAL: NCT01299883
Title: West Philadelphia Consortium to Address Disparities
Brief Title: West Philadelphia Consortium Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 5R24MDOO1594-06
Record Dates: First submitted 2011-02-01; First posted 2011-02-18 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Cancer; Cardiovascular Disease (CVD)
Keywords: Cancer; CVD; African American; Health Education Intervention; Intervention RCT; Study focus is to examine the influence of health education regarding either CVD or CVD and cancer on health behaviors.
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cancer and CVD Education (Active Comparator): Participants receive education about both cancer and CVD risk factors and their relationship to dietary and physical activity health behaviors.
  Interventions: Other: Integrated vs Non-integrated Risk Education
- CVD Education (Active Comparator): Participants receive education about CVD risk factors and their relationship to dietary and physical activity health behaviors.
  Interventions: Other: Integrated vs Non-integrated Risk Education

INTERVENTIONS:
Other: Integrated vs Non-integrated Risk Education — Integrated group receives education about risk factors for both cancer and CVD whereas the non-integrated group receives information about CVD only to assess differences in health behavior outcomes.

SUMMARY:
The investigators will evaluate the effects of an integrated risk counseling program on behavioral and psychological outcomes in African American men and women in a randomized trial that is implemented and evaluated collaboratively through the West Philadelphia Consortium to Address Disparities. The specific aims of this research are as follows:

1. To evaluate the effects of integrated versus disease specific counseling on risk exposure behaviors. The investigators predict that compared to individuals who receive disease specific counseling, those who receive integrated counseling will report greater intake of fruits and vegetables and increased rates of physical activity.
2. To evaluate effects of integrated versus disease specific counseling on psychological outcomes. The investigators predict that compared to individuals who receive disease specific counseling, those who receive integrated counseling will report greater risk comprehension related to cancer and cardiovascular disease and will be more motivated to make behavioral changes.
3. To identify the mechanisms through which integrated risk counseling leads to behavioral change. The investigators predict that changes in risk exposure behaviors (e.g., diet and physical activity) will be mediated by increased risk comprehension and self-efficacy for diet and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Age 18-75
* Resident of Philadelphia

Exclusion Criteria:

* Previous or current cancer diagnosis
* Previous or current diagnosis of a CVD
* Cognitive disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2008-08; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Dietary and physical activity behaviors | 12 months

SECONDARY OUTCOMES:
Exposure to program in terms of attendance | 4 wks.

CONTACTS AND LOCATIONS:
Overall Officials: Chanita H Halbert, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Community Based Research and Health Disparities, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Halbert CH, Bellamy S, Bowman M, Briggs V, Delmoor E, Purnell J, Rogers R, Weathers B, Kumanyika S. Effects of integrated risk counseling for cancer and cardiovascular disease in African Americans. J Natl Med Assoc. 2010 May;102(5):396-402. doi: 10.1016/s0027-9684(15)30574-5. PMID 20533774
- [Result] Halbert CH, Kumanyika S, Bowman M, Bellamy SL, Briggs V, Brown S, Bryant B, Delmoor E, Johnson JC, Purnell J, Rogers R, Weathers B. Participation rates and representativeness of African Americans recruited to a health promotion program. Health Educ Res. 2010 Feb;25(1):6-13. doi: 10.1093/her/cyp057. Epub 2009 Oct 29. PMID 19875730
- [Result] Weathers B, Barg FK, Bowman M, Briggs V, Delmoor E, Kumanyika S, Johnson JC, Purnell J, Rogers R, Halbert CH. Using a mixed-methods approach to identify health concerns in an African American community. Am J Public Health. 2011 Nov;101(11):2087-92. doi: 10.2105/AJPH.2010.191775. Epub 2011 Feb 17. PMID 21330592
- [Derived] Halbert CH, Bellamy S, Briggs V, Delmoor E, Purnell J, Rogers R, Weathers B, Johnson JC. A comparative effectiveness education trial for lifestyle health behavior change in African Americans. Health Educ Res. 2017 Jun 1;32(3):207-218. doi: 10.1093/her/cyx039. PMID 28335038